CLINICAL TRIAL: NCT06848725
Title: Testing the Implementation of a Toolbox to Optimize Data Collection and Data Quality of the National Medical Quality Indicators in Long-term Care Facilities: a Pilot Study Within the National Implementation Programme NIP-Q-UPGRADE
Brief Title: Testing the Implementation of a Toolbox to Optimize Data Collection and Data Quality of the National Medical Quality Indicators in Long-term Care Facilities: a Pilot Study. (NIP-Q-UPGRADE Subaim 1.8)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University of Applied Sciences and Arts of Southern Switzerland (Other); Institut et Haute Ecole de la Santé la Source (Other)
Responsible Party: Principal Investigator, Franziska Zúñiga, Prof. Dr. Franziska Zúñiga, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NIP-Q-UPGRADE WP 1.8
Record Dates: First submitted 2025-01-03; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Toolbox to Optimize Data Quality of the National MQIs
Keywords: NIP-Q-UPGRADE; quality indicators; long-term care; data quality improvement

STUDY DESIGN:
Intervention Model Description: The study addresses long-term care facilities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long-term care facilities (Experimental): All participating facilities will be offered the same toolbox
  Interventions: Behavioral: Data quality development toolkit concerning the medical quality indicators (MQI)

INTERVENTIONS:
Behavioral: Data quality development toolkit concerning the medical quality indicators (MQI) — The toolkit uses a train-the-trainer strategy.
  The research team will:
  * develop training and support materials for external training providers and delegated staff (champions) from the long-term care facilities
  * prepare external training providers within a one 3h session to train champions from the long-term care facilities
  * organize an e-mail contact centre for MQI related questions for the participating facilities.
  The external training providers will:
  - train the champions in one full day (8h) in-person training session and in 2 online sessions a 4h and 2h to support their co-workers to collect reliable MQI data.
  Based on the received training, the champions will:
  * provide internal trainings to the care and nursing team,
  * perform data quality monitoring,
  * provide feedback on data quality and act as a contact person for questions on MQI in their facility.

SUMMARY:
Since 2019, long-term care facilities in Switzerland are obliged by the Federal Insurance Law (KVG, Art. 59a) to report data for the calculation and public reporting of medical quality indicators (MQI). By 2024, this is done in four clinical domains: polypharmacy, pain, malnutrition and the use of physical restraints. This data is used for both monitoring quality of care on a national level and for internal quality of care development. To be valid and reliable, MQI data needs to be collected according to specified measurement instructions. An ethnographic study conducted within the NIP-Q-UPGRADE identified numerous challenges, which can lead to poor data quality.

The overall aim of this pilot study is to test the implementation of a data quality development toolkit concerning the MQI.

The toolkit uses a train-the-trainer strategy. The research team will prepare external training providers to train delegated staff from the long-term care facilities (further called champions), who will then train and support their co-workers to collect reliable MQI data. The research team developed training and support materials and organized an e-mail contact centre for MQI related questions for the participating facilities.

Implementation outcomes will be assessed at two levels: long-term care facilities and the external training providers.

Objectives at the external training provider level:

1. To determine the acceptability and feasibility of the training and support materials.
2. To determine the fidelity to the training and adaptations made when implementing it.
3. To identify the barriers and facilitators for the implementation of the training.
4. To measure the costs associated with delivering the training.

Objectives at the long-term care facility level:

1. To determine the acceptability and the feasibility of the data quality development toolkit components.
2. To determine the fidelity to toolkit components and adaptations made when implementing it.
3. To identify the barriers and facilitators for the implementation of the toolkit.
4. To measure the costs associated with implementing the toolkit.

DETAILED DESCRIPTION:
A one-group experimental study will be performed including a multiple methods evaluation.

Participants will be recruited at two levels:

* the provider responsible for delivering the training to the champions from the long-term care facilities,
* long-term care facilities who will implement the data quality development toolkit and select the champions to be sent to the training.

The external training provider is a company with experience in training staff of long-term care facilities in performing needs assessment with residents and in understanding and using the current MQI. The company will nominate employees to be instructed by the research team (December 2024) on how to conduct the developed training for facility champions. They will take up the organization and conduct of the trainings in three languages all regions of Switzerland. The research team will inform the training participants about the study and the data collection.

At facility level, five to ten long-term care facilities per Swiss language region (German, French and Italian speaking) will be recruited between November and December 2024 to implement the data quality development toolkit (i.e., a max. of 30 facilities in total over all language regions). At least one person per facility will be trained between January and March 2025 to act as a champion in the data quality development toolkit and perform tasks such as training of fellow staff and data quality monitoring (1 full day training onsite, two online trainings of 4h, resp. 2h with 2-4 weeks in-between). Trainings will be language-specific.

Individual study participants will be persons involved in delivering and coordinating champion trainings. In long-term care facilities we aim to collect data from the champions, the direct care staff at different educational levels, management staff and staff responsible for quality in the facilities. All individual participants will be asked to consent for data collection.

Data will be collected between November 2024 and June 2025:

At the training provider level

Quantitative data:

Activity logs: The costs of organizing and delivering the trainings will be assessed by using activity logbooks filled in continuously by the staff organizing and conducting the training (November to March 2025)

Qualitative data:

Interviews or group discussion: Acceptability, feasibility, fidelity, and adaptations to the toolkit, and barriers and facilitators to the implementation of the champion training will be assessed through interviews or group discussions with the involved staff after each of the three training session (January to March 2025, in total 9 interviews or group discussions, 3 per language region).

At the long-term care facility level

Quantitative data:

Online survey: Acceptability, feasibility and fidelity will be assessed via online surveys of involved staff at different levels (e.g., nurses, nurse assistants, management, champions) in March 2025. The surveys will also ask for background information on the facilities and participants.

Survey data will be collected in a secure online electronic data collection platform (REDCap).

Activity logbooks: Costs associated with the implementation will be assessed by using activity logbooks filled in by the champions and management.

Qualitative data:

Focus groups: Acceptability, feasibility, fidelity, and adaptations to the toolkit, and barriers and facilitators to implementation will be assessed through focus group per language region per staff group coming from different facilities:

1. 1-2 focus groups with management staff and staff responsible for quality (March 2025, total over all language regions 3-6 focus groups).
2. 1-2 focus groups with champions (March 2025 and June 2025, over all language regions 3-6 focus groups per time point, 6-12 in total)
3. 1-2 focus groups with nurses and care staff exposed to the toolkit (March 2025, total over all language regions 3-6 focus groups)

ELIGIBILITY:
Inclusion criteria:

1. External training providers:

   1. willing to implement trainings as designed by the research team and to all interested long-term care facilities
   2. have capacity to provide the trainers and infrastructure for the trainings - agree to non-commercial use of training materials
2. Trainer:

   1. with competence in training staff of long-term care facilities
   2. with knowledge on data collection of the current MQIs
3. Long-term care facilities:

   1. with a cantonal recognition as a residential long-term care facility
   2. willing to implement the toolkit
   3. which can nominate at least one champion
4. Champions:

   1. Long-term care facility employees motivated to take up the role
   2. having sufficient knowledge of the residents, infrastructure and processes in the facility (e.g., resident care, needs assessment instrument, electronic health records)
   3. Ideally with experience in leadership, staff training, MQI data collection and quality monitoring, e.g., nurse, nurse expert, quality manager, needs assessment instrument manager
5. Management and staff responsible for quality:

   1. any level of management staff and staff responsible for quality in long-term care facility e.g., director of nursing, team leader, quality manager
   2. directly involved in supporting the implementation of the toolkit or exposed to its content
6. Nursing and care staff:

   1. Any level of nursing or care staff e.g., registered nurses, licensed practical nurses, nurse aids involved in collecting data for MQI
   2. exposed to the content of the toolkit (i.e., internal trainings, feedback, support materials), e.g., registered nurses, licensed practical nurses, nurse aids

Exclusion criteria:

1. long-term care facilities that are participants of the study "Data Quality and National Quality Indicators in Long-term Care Facilities: a Validation Study and Evaluation Study"

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the toolbox | After each champion's training unit (baseline, 3 weeks and 9 weeks): interview with trainer. At 3 months: survey and focus groups with champions, leadership, nursing and care staff. At 6 months: focus group with champions.
  Acceptability of toolbox components will be assessed in a survey with Acceptability of Intervention Measure (AIM), a 4-item instrument measuring the acceptability of an intervention.
  Further exploration of acceptability in qualitative interviews and focus groups
Feasibility of the toolbox | After each champion's training unit (baseline, 3 weeks and 9 weeks): interview with trainer. At 3 months: survey and focus groups with champions, leadership, nursing and care staff. At 6 months: focus group with champions.
  Feasibility of toolbox components will be assessed in a survey with Feasibility of Intervention Measure (FIM), a 4-item instrument measuring the feasibility of an intervention.
  Further exploration of feasibility in qualitative interviews and focus groups.
Implementation fidelity | After each champion's training unit (baseline, 3 weeks and 9 weeks): interview with trainer. At 3 months: survey and focus groups with champions, leadership, nursing and care staff. At 6 months: focus group with champions.
  Degree of fidelity to each component (yes, partial, no) will be measured using a questionnaire survey.
  Further exploration of implementation fidelity in qualitative interviews and focus groups.
Barriers to the implementation of the toolbox | After each champion's training unit (baseline, 3 weeks and 9 weeks): interview with trainer. At 3 months: focus groups with champions, leadership, nursing and care staff. At 6 months: focus group with champions.
  Barriers to the implementation will be explored in qualitative interviews and focus groups, and categorized according to the Consolidated Framework of Implementation Research (CFIR)
Facilitators to the implementation of the toolbox | At 3 months: focus groups with champions, leadership, nursing and care staff. At 6 months: focus group with champions.
  Facilitators to the implementation will be explored in qualitative interviews and focus groups, and categorized according to the Consolidated Framework of Implementation Research (CFIR)
Sum of costs associated with implementation of the toolkit in Swiss francs | Continuously from baseline training to 3 months after
  Costs will be calculated based on time spent on implementation activities per staff group with corresponding hourly salary estimate, recorded in an activity logbook

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Zúñiga, Prof. Dr., Principal Investigator — University of Basel
Locations (3):
- Switzerland (3):
  - Department of Business Economics, Health and Social Care, University of Applied Sciences and Arts of Southern Switzerland (SUPSI), Manno, Switzerland., Manno, Canton Ticino
  - Institut für Pflegewissenschaft - Nursing Science (INS), University of Basel, Basel
  - La Source School of Nursing, HES-SO University of Applied Sciences and Arts of Western Switzerland, Lausanne, Switzerland, Lausanne

IPD SHARING:
Plan to Share IPD: No